CLINICAL TRIAL: NCT03609931
Title: Patient Specific Mitral Valve Modeling for Surgical Planning and Training
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Responsible Party: Principal Investigator, Daniel Bainbridge, Associate Professor, London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's
Other Study IDs: 111462
Record Dates: First submitted 2018-06-12; First posted 2018-08-01 (Actual); Last update posted 2018-08-01 (Actual); Status verified 2018-07

CONDITIONS: Mitral Valve Prolapse; Mitral Regurgitation; Mitral Valve Disease
Keywords: Mitral Valve
MeSH Terms: conditions — Mitral Valve Prolapse; Mitral Valve Insufficiency

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Mitral Valve repair: Patients undergoing mitral valve repair
  Interventions: Procedure: Mitral Valve Model

INTERVENTIONS:
Procedure: Mitral Valve Model — Creation of a mitral valve patient specific model to see if it mimics the patients valve

SUMMARY:
Mitral valve disease is a common pathologic problem occurring in approximately 2% of the general population but climbing to 10% in those over the age of 75 in Canada[1]. This project has three primary goals all of which will positively affect cardiac patient care.

1) Create patient specific MV models for complex repairs that will allow surgeons the opportunity to practice the repair. 2) Potentially predict the outcomes following minimally invasive repair techniques such as transcatheter treatments (e.g., MitraClip). 3) Provide a model to train individuals on mitral valve repair techniques.

DETAILED DESCRIPTION:
BACKGROUND Mitral valve disease is a common pathologic problem occurring in approximately 2% of the general population, but climbing to 10% in those over the age of 75 in Canada. Of this group, approximately 20% have a sufficiently severe form of the disease that may require surgical intervention to restore normal valve function and prevent early mortality [4]. Evidence indicates that the surgeon's individual volume of mitral valve repair cases performed is a determinant of not only successful mitral repair rates, but also freedom from reoperation, and patient survival. For patients previously deemed inoperable due to co-morbidities, new techniques to treat mitral valve disease are being developed. However, assessing the optimal approach and the point at which clinical benefit is exceeded by the poor value or futility of the procedure is one of the biggest clinical challenges for physicians.

In the past decade, 3D echocardiography has emerged as a standard of care in diagnostic and interventional imaging for cardiac surgery and cardiology. This, coupled with the emergence of inexpensive 3D printing technology has led researchers and clinicians to explore how improved imaging and additive manufacturing can be used to improve patient outcomes.

In this context, the investigators have completed a proof-of-concept workflow for creating dynamic, patient specific mitral valve models. In concert with a left ventricle simulator 8], these valve models can mimic patient valve pathologies both anatomically and dynamically, as shown in Doppler ultrasound. In a 10 patient retrospective study, the investigators have demonstrated the ability to accurately re-create patient pathology, perform realistic surgical repairs, and assess realistic valve function post repair. The study team's vision is to create a simulator that can be used to assess patient candidacy for percutaneous interventions, assess different repair options for both percutaneous and surgical interventions, and finally use the model as a simulator for competency-based MV interventions.

RATIONALE Based on our successful proof of concept, the goal is to translate this technology to clinical use by validating our valve models. There are two primary long term goals. First, to validate a system for using patient specific MV models to: 1- assess intervention options, and 2: plan repair strategies for improved patient outcomes. Second, by building a database of MV pathologies, create a competency based simulator/trainer to provide surgeons with increased experience in MV repair techniques.

OBJECTIVES

1. Validate the accuracy of patient specific MV pathologies and repairs in a prospective 65 patient study;
2. Optimize our work-flow for creating valve models, in terms of accuracy, manufacture time required, and expense;
3. Validate the accuracy of our patient models for both surgical cases and transcatheter MitraClip interventions;

ELIGIBILITY:
Inclusion Criteria:

* Patients undergo mitral valve repair with either surgery of MitraClip techniques
* Over 18 years old

Exclusion Criteria:

* Unable to place TEE probe
* Refuse consent

Ages: 18 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Adult patients with mitral regurgitation scheduled to undergo mitral valve repair with either a open heart surgical technique or with a MitraClip
Sampling Method: Non-Probability Sample
Enrollment: 65 (Estimated)
Dates: Start 2018-07 (Estimated); Primary Completion 2019-08 (Estimated); Study Completion 2020-01 (Estimated)

PRIMARY OUTCOMES:
MR following patient/model repair | Creation and assessment of the model within 1 week before or after surgery/intervention on the patient.
  The degree and location of residual MR following mitral repair surgery

SECONDARY OUTCOMES:
2D measurements of the mitral valve: Anterolateral-Posteromedial Diameter | Assessment of model within 1 week of surgical or interventional repair on the patient
  A 2D measurements taken from the echocardiography images of the mitral valve and model
2D measurements of the mitral valve:Annular Height | Assessment of model within 1 week of surgical or interventional repair on the patient
  A 2D measurements taken from the echocardiography images of the mitral valve and model
2D measurements of the mitral valve: Annular 3D Circumference | Assessment of model within 1 week of surgical or interventional repair on the patient
  A 2D measurements taken from the echocardiography images of the mitral valve and model
2D measurements of the mitral valve:Annular 2D Area | Assessment of model within 1 week of surgical or interventional repair on the patient
  A 2D measurements taken from the echocardiography images of the mitral valve and model
2D measurements of the mitral valve: Annular Ellipticity | Assessment of model within 1 week of surgical or interventional repair on the patient
  A 2D measurements taken from the echocardiography images of the mitral valve and model
2D measurements of the mitral valve: Anterior Leaflet 3D Area | Assessment of model within 1 week of surgical or interventional repair on the patient
  A 2D measurements taken from the echocardiography images of the mitral valve and model
2D measurements of the mitral valve: Posterior Leaflet 3D Area | Assessment of model within 1 week of surgical or interventional repair on the patient
  A 2D measurements taken from the echocardiography images of the mitral valve and model
2D measurements of the mitral valve: Leaflet 3D Area | Assessment of model within 1 week of surgical or interventional repair on the patient
  A 2D measurements taken from the echocardiography images of the mitral valve and model
2D measurements of the mitral valve: Mitral Regurgitation Orifice Area | Assessment of model within 1 week of surgical or interventional repair on the patient
  A 2D measurements taken from the echocardiography images of the mitral valve and model
2D measurements of the mitral valve: Tenting Volume | Assessment of model within 1 week of surgical or interventional repair on the patient
  A 2D measurements taken from the echocardiography images of the mitral valve and model
2D measurements of the mitral valve: Nonplanar Angle | Assessment of model within 1 week of surgical or interventional repair on the patient
  A 2D measurements taken from the echocardiography images of the mitral valve and model
2D measurements of the mitral valve: tenting Height. | Assessment of model within 1 week of surgical or interventional repair on the patient
  A 2D measurements taken from the echocardiography images of the mitral valve and model
ICU LOS | Postoperative period until ICU discharge (expected mean of 1 days)]
  length of stay in the ICU
Hospital LOS | Postoperative period until hospital discharge (expected mean of 5 days)
  Length of stay in hospital
Delirium | Postoperative period until hospital discharge (expected mean of 5 days)
  Delirium in hospital
Renal failure requiring dialysis | Postoperative period until hospital discharge (expected mean of 5 days)
  Dialysis
Stroke,TIA | Postoperative period until hospital discharge (expected mean of 5 days)
  Diagnosis of stroke
Death in Hospital | Postoperative period until hospital discharge (expected mean of 5 days)
  Death
Reoperation for Bleeding | Postoperative period until hospital discharge (expected mean of 5 days)
  Return to the operating room for re-exploration of the surgical procedure due to excess blood loss in the ICU

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ginty O, Moore J, Peters T, Bainbridge D. Modeling Patient-Specific Deformable Mitral Valves. J Cardiothorac Vasc Anesth. 2018 Jun;32(3):1368-1373. doi: 10.1053/j.jvca.2017.09.005. Epub 2017 Sep 7. PMID 29221976